CLINICAL TRIAL: NCT05790655
Title: Ovarian Platelet-Rich Plasma Injections for Diminished Ovarian Reserve Patients: A Double-Blinded Placebo-Control Trial
Brief Title: Ovarian PRP for Diminished Ovarian Reserve
Acronym: oPRP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Generation Next Fertility (Other)
Collaborators: Igenomix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IORG0010499_202301
Record Dates: First submitted 2023-03-06; First posted 2023-03-30 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Diminished Ovarian Reserve
Keywords: Ovarian Platelet Rich Plasma; DOR; Ovarian PRP; IVF; PRP; PGT-A; ICSI

STUDY DESIGN:
Intervention Model Description: Prospective, double-blinded placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient and PI will not know which arm the patient is in. This will not be unblinded until study completion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oPRP injections (Experimental): Patients own prepared PRP will be injected into each ovary
  Interventions: Other: oPRP
- Placebo (Placebo Comparator): Patient's serum will be injected into the ovary (not rich with platelets)
  Interventions: Other: Placebo- Serum

INTERVENTIONS:
Other: oPRP — Prepared sample from patient's own blood collected and processed. Either PRP or serum is injected into the patient's ovary. All other care is standard for the IVF process
  Arms: oPRP injections
Other: Placebo- Serum — Patient's serum is injected into ovary instead of PRP as placebo
  Arms: Placebo

SUMMARY:
This prospective double-blinded randomized placebo control study aims to determine if In Vitro Fertilization (IVF) outcomes are improved by ovarian platelet-rich plasma injections (oPRP) for women diagnosed with diminished ovarian reserve (DOR). Women with DOR notoriously have the lowest chance of pregnancy and live birth compared to age-matched peers with a normal or robust ovarian reserve.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled trial comparing ovarian injection of platelet-rich plasma vs. placebo in women diagnosed with diminished ovarian reserve at risk for a poor ovarian response (POR) between 35 to 42 years of age. Participants for this study include patients who are planning to undergo IVF with preimplantation genetic testing for aneuploidy (PGT-A) followed by a frozen embryo transfer (FET) cycle. Only patients with either a euploid embryo or eligible mosaic embryo (following consultation with a geneticist), as determined by PGT-A, will be allowed to proceed with a single blastocyst FET cycle

All patients will have a baseline ultrasound and blood work at the time of menses, approximately one month prior to starting their initial IVF cycle. Routine monitoring will be required to determine the day of ovulation. Once an LH surge is detected or if a lead follicle on pelvic ultrasound is deemed large enough to induce ovulation, a "trigger" shot with 250 mcg/0.5 mL of Ovidrel® will be self-administered subcutaneously (SQ). Based upon the patient's randomization, either oPRP or ovarian Serum (oS) injections will be performed under anesthesia and within 72 hours from the day of ovulation. Following their ovarian injections, all patients will return for monitoring with the onset of menses approximately 14 to 16 days from the date of ovulation.

A medication protocol will be determined at the start of each IVF cycle. Either a natural (nIVF), mild (mIVF) or conventional (cIVF) IVF protocol will be chosen by the treating physician. This determination will be based on findings from the repeat pelvic ultrasound with AFC and blood work for anti-mullerian hormone (AMH), follicle stimulating hormone (FSH), lutenizing hormone (LH), estradiol (E2), progesterone (P4), and beta-human chorionic gonadotrophin (B-hCG). Natural IVF will be considered for patients with only 1-2 antral follicles, mIVF for patients with 2-4 antral follicles observed, and cIVF for patients with four or more antral follicles visualized at the time stimulation started.

Patients will begin their designated protocol and return four to five days following medication start. A repeat pelvic ultrasound will be performed to measure the growth and size of all follicles visualized along with the endometrial thickness. Also, blood work for E2, FSH, LH, and P4 will be obtained. Monitoring for follicular and endometrial development will continue routinely and as needed, until the majority of all follicles observed have a mean diameter between 15 to 22 mm. Induction of ovulation will commence 35 and a half hours prior to oocyte retrieval, by self-administration of 10,000 IU hCG SQ.

The patient will receive deep IV sedation anesthesia by a board-certified anesthesiologist for her oocyte retrieval and placement of either her second oPRP or oS injections. Using transvaginal ultrasound guidance, all follicles visualized under ultrasound will be aspirated using standard practices by patients undergoing IVF at GNF. Aspirates will be collected in 10 ml test tubes. All oocytes will be assessed at the time of retrieval for maturity. All oocytes that are deemed mature (MII) will undergo intracytoplasmic sperm injection (ICSI), to maximize fertilization rates, 2-4 hours after identification of the first polar body. All immature (non MII) oocytes will be isolated under a stereomicroscope and transferred into maturation media and incubated further in a triple gas mixture (90% N2, 5% CO2, and 5% O2) for up to 24 hours to allow maturation prior to ICSI. Following the oocyte retrieval, either oPRP or oS will be performed as described previously.

Monitoring will recommence two weeks following the first oocyte retrieval to identify if any residual follicles or ovarian cysts are present. If the ovaries are deemed resting and no active ovarian cysts persist, then the patient will begin her second IVF cycle. Again, the medication protocol will be determined by findings observed on pelvic ultrasound including AFC and ovarian hormone testing. If the patient is deemed ineligible to start another IVF cycle, then she will return with the following menstrual period to begin her second IVF cycle. The process of monitoring patients, inducing ovulation and collecting oocytes will be identical to the first oocyte retrieval. However, no additional oPRP or oS injections will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of diminished ovarian reserve
* Clinical diagnosis of poor ovarian response
* Women age 35-42

Exclusion Criteria:

* Clinical diagnosis of premature ovarian failure
* Clinical diagnosis of menopause.
* Under 35 years of age
* Over 42 years of age

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-10-07 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
oPRP changes Ovarian Response and the total Number of oocytes retrieved | 12 months
  Total oocyte yield
oPRP impacts the Number or Euploid Embryos available for frozen embryo transfers | 12 months
  Available embryos for frozen embryo transfers

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Hade, MD, Principal Investigator — Generation Next Fertility
Locations (1):
- Generation Next Fertility, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Collaboration to share protocol may be requested with PI
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: April 2023 to April 2024
Access Criteria: Protocol may be shared with other research bodies upon request for collaboration
URL: http://www.generationnextfertility.com

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT05790655/Prot_ICF_000.pdf